CLINICAL TRIAL: NCT01339455
Title: Autologous Hematopoietic Stem Cell Transplant in Patients With Neuromyelitis Optica
Brief Title: Autologous Hematopoietic Stem Cell Transplant in Neuromyelitis Optica
Acronym: SCT-NMO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: recruitment failure
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Jodie Burton MD, MSc, FRCPC, Assistant Professor, University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHREB ID# 23282
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Neuromyelitis Optica
Keywords: Neuromyelitis Optica; NMO; Devic's Disease; Stem Cell Transplant
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AHSCT (Experimental): All patients undergo autologous hematopoietic stem cell transplantation in a two stage process.
  Interventions: Procedure: AHSCT

INTERVENTIONS:
Procedure: AHSCT — AHSCT Procedure:
  1. Mobilization and Harvesting:
     * Cyclophosphamide
     * Rituximab
     * GSCF
     * Dexamethasone
     * Apheresis
  2. Conditioning and Infusion (3-4 weeks after Mobilization and Harvesting):
     * Cyclophosphamide
     * MESNA
     * Rabbit ATG
     * Rituximab
     * Methylprednisolone
     * Stem Cell infusion
     * GSCF

SUMMARY:
Neuromyelitis Optica (NMO) is a demyelinating and degenerative disorder of the CNS affecting vision and spinal cord function. This disease is rare compared to Multiple Sclerosis (MS), but it is devastating and often leads to accumulating disability with a 5 year-mortality of approximately 30%. Survivors are typically left with severe morbidity secondary to blindness, quadriparesis and respiratory failure. No agent has been found to be highly effective in halting disease activity. Based on recent outcomes of stem cell transplant trials and reports in autoimmune diseases including MS, and based on the mechanisms of NMO, we anticipate that stem cell transplantation may provide lasting disease stability for NMO patients. The hypothesis of the present trial is that autologous hematopoetic stem cell transplantation in patients with NMO will provide lasting benefit in relapse prevention. Specifically, we anticipate a 50% reduction in the proportion of patients experiencing relapse over a three year period. We will be following patients for a total of five years after transplantation.

DETAILED DESCRIPTION:
Patients who are deemed eligible will be enrolled and undergo a two stage transplant process followed by neurological assessments every 6 months for the following 5 years assessing EDSS, visual metrics, MRI, AQP-4 antibodies, MSFC and SF36.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65, inclusive
* Diagnosis of NMO using Wingerchuk 2006 NMO Criteria
* EDSS 0-6.5
* Treatment with a minimum of one NMO therapy in past 12 months
* One objective and documented relapse in the past 12 months and two relapse events in the past 24 months despite medical therapy
* ECOG performance status 0-3
* Platelets ≥100 x 109/L
* ALT ≤3 x ULN
* Total bilirubin ≤2.0 x ULN, except in patients with Gilbert syndrome or in patients in whom the bilirubin rise is of non-hepatic origin
* Serum creatinine <1.5 x ULN or creatinine clearance ≥50 cc/min
* Patients must reside in Alberta, Canada for the duration of the transplant period of the trial

Exclusion Criteria:

* Any illness that would jeopardize the ability of the patient to complete study protocol
* Prior malignancy unless non-melanoma skin cancer, carcinoma in-situ of the cervix (CIN) or breast, or malignancy treated more than 5 years previously with no evidence of recurrent disease since initial treatment
* Pregnant or lactating females. Women of childbearing potential must have a negative serum or urine β-hCG pregnancy test at screening
* Inability or unwillingness to pursue effective means of birth control
* FEV1/FVC < 50% of predicted
* DLCO < 50% of predicted
* Resting LVEF < 50 %
* Known hypersensitivity to mouse, rabbit, or E. Coli derived proteins, or to iron compounds/medications
* Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams
* Unable or unwilling to provide written informed consent for participation
* Active infection except asymptomatic bacteriuria
* Any use of investigational therapies within 4 weeks prior to initiation of study treatment
* Patients dependent on prednisone who cannot be successfully tapered to a maximum of 0.5mg/kg/d prior to mobilization therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Proportion relapse-free at three years | 3 years
  The proportion of surviving patients who are relapse-free at three years after transplant

SECONDARY OUTCOMES:
Proportion relapse-free at five years | 5 years
  The proportion of surviving patients relapse-free at year five
Relapse count | Annually over 5 years
  Number of NMO relapse events
Disability progression | Over 5 years
  Time to progression of EDSS by one step
Retinal nerve fiber layer (RFNL) status | 5 years
  Change in RNFL by optical coherence tomography over trial
25 foot timed walk test | 5 years
  Change in 25 ft timed walk test over trial
PASAT | Annually over 5 years
  Annual and change from baseline to end of trial in Paced Auditory Serial Addition Test to assess cognitive function.
Hospitalization | Over 5 years
  Number of hospitalizations, days in hospital over trial period
Overall survival | Over 5 years
  Survival over trial period
Time to next relapse | Over 5 years
  Time to next relapse after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jodie M Burton, MD,MSc,FRCPC, Principal Investigator — Department of Clinical Neurosciences, Hotchkiss Brain Institute, University of Calgary; Jan Storek, MD,PhD, Principal Investigator — Department of Medicine, University of Calgary
Locations (1):
- Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada